CLINICAL TRIAL: NCT04823715
Title: Transarterial Chemoembolization Plus Hypofractionnated Radiotherapy vs. Surgery in Locally Advanced Hepatocellular Carcinoma: an IPTW Comparison
Acronym: TACE-hypoRT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 249
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Non-metastatic Hepatocellular Carcinoma
Keywords: Liver neoplasms; Carcinoma; Hepatocellular; Radiation therapy; TACE; Transarterial Chemoembolization
MeSH Terms: conditions — Liver Neoplasms; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TACE- hypofractionated radiation therapy: Patients will receive one course of transarterial chemoembolization followed 1 to 4 weeks later by hypofractionated radiation therapy up to a total dose of 45 to 60 Gy, 3 Gy per fraction, 5 fractions per week, for an overall treatment time of 3 to 4 weeks.
  Interventions: Other: TACE + hypofractionated EBRT
- Surgical resection: Surgical resection by open-laparotomy or laparoscopy of hepatocellular carcinoma
  Interventions: Procedure: Surgical resection

INTERVENTIONS:
Other: TACE + hypofractionated EBRT — One cure of doxorubicin or DC Beads transarterial chemoembolization by a highly experienced interventional radiologist, followed 1 to 4 weeks later by hypofractionated external beam radiation therapy up to a total dose of 45-60 Gy, 3 Gy per fraction, 5 fractions per week, for an overall treatment time of 3 to 4 weeks.
  Groups: TACE- hypofractionated radiation therapy
Procedure: Surgical resection — Surgical resection by open-laparotomy or laparoscopy of hepatocellular carcinoma by a highly experienced liver surgeon
  Groups: Surgical resection

SUMMARY:
Patients with non-metastatic unresectable hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age
* ECOG 0-2
* Histologically proven hepatocellular carcinoma or proven according to radiological and biochemical criteria (EASL-AASLD) in cirrhotic patients
* Child-Pugh class A
* Absence of truncular or lobar portal vein invasion, or suprahepatic vein invasion

Exclusion Criteria:

* Uncontrolled replication of hepatitis B virus
* Transplanted liver
* Previous abdominal irradiation
* Previous treatment of HCC with systemic therapy, or with surgical resection in the 2 previous years
* Metastatic illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 or older, presenting Child-Pugh class A HCC treated in Hospices Civils de Lyon between 2004 and 2016
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Disease-free survival of the patient after start of treatment | Within 10 years after the treatment (surgical resection or TACE)
  Disease-Free Survival (DFS) defined as the time (in months) between the treatment (surgical resection or TACE) and the diagnostic of local, locoregional or distant recurrence, or date of death from any cause; patients who are alive or lost to follow-up at the time of the analysis will be censored on the last follow-up date; patients who have received a liver transplant for non-carcinologic reason will be censored on the date of transplantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon, France